CLINICAL TRIAL: NCT04104295
Title: The Use of Ultrasound to Determine Correct Nasogastric Tube Placement in Children Admitted to the Pediatric ICU: a Pilot Study
Brief Title: The Use of Ultrasound in Nasogastric Tube Placement in Children Admitted to the Pediatric ICU
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Study never began.
Sponsor: Yale University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2000026488
Record Dates: First submitted 2019-09-24; First posted 2019-09-26 (Actual); Last update posted 2021-04-20 (Actual); Status verified 2021-04

CONDITIONS: Nasogastric Tube
Keywords: nasogastric tube; ultrasound
MeSH Terms: interventions — Ultrasonography

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Ultrasound following X-ray (Experimental): An ultrasound scan of the abdomen within 2 hours of the routine X-ray will be performed by a physician blinded to the X-ray results.
  Interventions: Diagnostic Test: Ultrasound following X-ray

INTERVENTIONS:
Diagnostic Test: Ultrasound following X-ray — A short (less than 10 minutes) ultrasound (US) scan of the abdomen within 2 hours of the routine X-ray (XR). The performer will be a physician who received a focused training on relevant US views, blinded to the XR image and report.
  Other Names: Ultrasound

SUMMARY:
The purpose of this study is to determine if ultrasound (US), when used by the clinician, can determine the presence of nasogastric tube (NGT) in the stomach of patients admitted to the pediatric intensive care unit (PICU).

DETAILED DESCRIPTION:
Currently, the standard of care is to routinely obtain an X-ray (XR) after every nasogastric tube (NGT) placement in the pediatric intensive care unit (PICU). After obtaining informed consent and the child's assent, a short (less than 10 minutes) ultrasound (US) scan of the abdomen within 2 hours of the routine XR.

ELIGIBILITY:
Inclusion Criteria:

* PICU patient undergoing routine NGT insertion by nursing staff

Exclusion Criteria:

* Any contraindication for US probe placement such as skin infection and abdominal wounds.
* Hemodynamically unstable patients.
* Patients for whom NGT placement will not be verified by XR, such as Ataxia Telangiectasia patients.

Ages: 0 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 0 (Actual)
Dates: Start 2020-03-24 (Estimated); Primary Completion 2020-09-30 (Estimated); Study Completion 2021-01-31 (Estimated)

PRIMARY OUTCOMES:
Correct placement of NG tube | Up to 10 minutes
  The operational definition will be the number of correct identification of NG tube position using ultrasound, as compared to the official X-ray read.

CONTACTS AND LOCATIONS:
Overall Officials: Eitan Neeman, MD, Principal Investigator — Yale University - MEDPED Critical Care

IPD SHARING:
Plan to Share IPD: No